CLINICAL TRIAL: NCT01108289
Title: The Oxytocin Initiative: Determining the Effect of Prophylactic Administration of Oxytocin in Uniject™ by a Community Health Officer on Postpartum Hemorrhage at Home Births in Four Districts in Ghana
Brief Title: Effect of Prophylactic Administration of Oxytocin in Uniject™ on Postpartum Hemorrhage at Home Births in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); PATH (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAT.1429-07882-1
Record Dates: First submitted 2010-04-02; First posted 2010-04-21 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Postpartum Hemorrhage
Keywords: hemorrhage; uterotonic; oxytocin; blood loss; community; Ghana; randomized trial
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin in Uniject (Experimental): Community Health Officers will provide 10 IU Oxytocin in Uniject device IM immediately after delivery of baby
  Interventions: Other: Oxytocin in Uniject
- PPH Treatment Only (No Intervention): Community Health Officers will be able to treat for PPH only, not provide Oxytocin in Uniject

INTERVENTIONS:
Other: Oxytocin in Uniject — 10 IU Oxytocin delivered intramuscularly immediately after delivery of the baby
  Other Names: uterotonic, pitocin
  Arms: Oxytocin in Uniject

SUMMARY:
This study is designed to test the hypothesis that the intramuscular administration of 10 IU of oxytocin in Uniject™ during the third stage of labor by a Community Health Officer (CHO) at home births in Ghana will reduce the risk of postpartum hemorrhage by 50 percent relative to home births attended by the same type of provider who does not provide a uterotonic drug.

ELIGIBILITY:
Inclusion Criteria:

* home delivery
* presence of Community Health Officer at time of delivery

Exclusion Criteria:

* None

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1586 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
postpartum hemorrhage-1 | after delivery of baby
  blood loss >=500 ml after delivery of the baby, as measured through plastic calibrated drape
postpartum hemorrhage-2 | after delivery of the baby
  blood loss >=500ml OR treatment dose of oxytocin provided
postpartum hemorrhage-3 | after delivery of the baby
  blood loss >=500ml OR treatment dose of oxytocin provided OR referral for bleeding

SECONDARY OUTCOMES:
Oxytocin use before delivery | labor and delivery
  the proportion of deliveries where oxytocin in uniject was administered prior to the delivery of the baby
stillbirth | labor/delivery
  stillbirth is defined as death of a fetus after 28 weeks of gestation, prior to birth
neonatal death | first month of life
  neonatal death is defined as death of a live born baby prior to completion of 28 days
need for neonatal resuscitation | 0-6 hours after birth

OTHER OUTCOMES:
Postpartum Hemorrhage >=1000ml | after delivery of the baby
  1000ml or more blood is observed in the collection drape

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stanton, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Sam Newton, MD, PhD, Principal Investigator — Kintampo Health Research Center, Kintampo, Ghana
Locations (1):
- Kintampo Health Research Center, Kintampo, Brong Ahafo, Ghana

REFERENCES:
- [Derived] Stanton CK, Newton S, Mullany LC, Cofie P, Tawiah Agyemang C, Adiibokah E, Amenga-Etego S, Darcy N, Khan S, Armbruster D, Gyapong J, Owusu-Agyei S. Effect on postpartum hemorrhage of prophylactic oxytocin (10 IU) by injection by community health officers in Ghana: a community-based, cluster-randomized trial. PLoS Med. 2013 Oct;10(10):e1001524. doi: 10.1371/journal.pmed.1001524. Epub 2013 Oct 1. PMID 24130463
- [Derived] Stanton CK, Newton S, Mullany LC, Cofie P, Agyemang CT, Adiibokah E, Darcy N, Khan S, Levisay A, Gyapong J, Armbruster D, Owusu-Agyei S. Impact on postpartum hemorrhage of prophylactic administration of oxytocin 10 IU via Uniject by peripheral health care providers at home births: design of a community-based cluster-randomized trial. BMC Pregnancy Childbirth. 2012 Jun 7;12:42. doi: 10.1186/1471-2393-12-42. PMID 22676921